CLINICAL TRIAL: NCT03585491
Title: Shoulder Instability Trial Comparing Arthroscopic Stabilization Benefits Compared With Latarjet Procedure Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moin Khan (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other); University of Western Ontario, Canada (Other); The Ottawa Hospital (Other); Pan Am Clinic (Other); University of Colorado, Denver (Other); Queen's University (Other); Sunnybrook Health Sciences Centre (Other); Boston University (Other); Deventer Ziekenhuis (Other); Banff Sport Medicine Foundation (Other); McMaster University (Other); Brantford General Hospital (Unknown); London Health Sciences Centre (Other); Parc de Salut Mar (Other); Hospital Universitari de Bellvitge (Other); Hospital de Terrassa (Other); Hospital Mutua de Terrassa (Other); Pontificia Universidad Catolica de Chile (Other); Endeavor Health (Other); Medstar Health Research Institute (Other); Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor-Investigator, Moin Khan, MD, MSc, FRCSC, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STABLE
Record Dates: First submitted 2018-06-28; First posted 2018-07-13 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Dislocation; Sport Injuries; Shoulder; Anterior Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bankart + Remplissage Procedure (Experimental): Bankart Procedure: the participant will be placed in the lateral decubitus or beach chair position. Standard diagnostic arthroscopy will be performed. The anterior capsulolabral complex will be freed from the anterior aspect of the scapular neck. The anterior aspect of the scapular neck will be decorticated using a motorized burr. A capsuloligamentous repair will be performed with the capsule shifted from inferior to superior and repaired on the glenoid face. The number of anchors used for the repair will be left to the discretion of the surgeon. Patients will be given a sling for 4 weeks, and participation in sports will not be allowed for 6 months.
  Interventions: Procedure: Bankart + Remplissage Procedure
- Latarjet Procedure (Experimental): Open or Arthroscopic coracoid transfer (Latarjet Procedure): This procedure may be performed through small incisions (minimally invasive) but may require a larger incision in some cases. It involves the transfer of a nearby bony structure (the coracoid process) to the front of the shoulder joint (glenoid). This bone will then provide support to prevent the shoulder joint from dislocating.
  Interventions: Procedure: Latarjet Procedure

INTERVENTIONS:
Procedure: Latarjet Procedure — Participants will undergo open or arthroscopic Latarjet procedure.
  Arms: Latarjet Procedure
Procedure: Bankart + Remplissage Procedure — Participants will undergo arthroscopic stabilization.
  Arms: Bankart + Remplissage Procedure

SUMMARY:
The primary objective of the pilot study is to assess the feasibility of a definitive trial to determine the effect of arthroscopic capsuloligamentous repair (Bankart + Remplissage) vs. coracoid transfer (Latarjet procedure) on recurrent dislocation rates and functional outcomes over a 24-month period.

DETAILED DESCRIPTION:
Background:

Shoulder is a highly mobile joint with the most directional range of movement compared to other joints in the body. Thus, the surrounding supporting structures of the shoulder joint compromise on the stability of the joint, in order to accomplish this wide range of motion.

Anterior dislocations, the most common type of shoulder dislocation, are often complicated by instability, and repeated dislocations. Shoulder instability results in pain and negatively impacts quality of life. Several long-term studies have demonstrated a relationship between the repeated dislocations and the risk of arthritis.

Surgical stabilization of the shoulder improves function and may reduce the risk of developing degenerative arthritis. Two procedures are commonly performed in patients with repeated dislocations: a bony transfer procedure (Latarjet) or a soft tissue procedure (Bankart + Remplissage). The Latarjet procedure involves transferring bone to the front of the shoulder. The Bankart + Remplissage procedure involves tightening the soft tissues at the front of the shoulder joint.

Although retrospective clinical studies have suggested a reduced recurrence rate with the Latarjet procedure, there is a higher reported complication rate and potential morbidity associated with the open procedure. Several case series from high-volume surgeons in Europe have suggested the Latarjet repair to be an acceptable and potentially favorable surgical approach for all cases of recurrent anterior shoulder dislocation, even in the primary setting and in the absence of significant glenoid cup bone loss. Retrospective analysis of soft tissue repair in comparison to open coracoid (Latarjet) procedure found at 10-year follow up, redislocation rates were 13% (36) of 271 shoulders with a Bankart repair and 1% (1) of the 93 shoulders with a Latarjet repair.

Need for a Pilot Study Prior to a Large Trial:

No comparative randomized control trial has been completed evaluating Bankart repair in comparison to Latarjet procedure in the setting of mild to moderate bone loss. Thus, surgeons face uncertainty regarding which procedure to perform. The Latarjet is more invasive (larger incision) and some research suggests it may be more effective at treating instability. The Bankart procedure, while minimally invasive (smaller incision), may result in higher rates of instability after surgery.

Prior to a large trial, the investigators will conduct a pilot trial comparing arthroscopic capsuloligamentous repair (Bankart Procedure) vs. coracoid transfer (Latarjet procedure) on recurrent dislocation rates and functional outcomes over a 24-month period. This research will provide surgeons with new information regarding the best treatment for recurrent shoulder dislocation.

Study Aims and Objectives:

A pilot study is needed prior to a large trial to determine the feasibility of a larger trial in terms of:

1. Ability to recruit across clinical sites
2. Adherence to study protocol and,
3. Ability to follow participants for 24 months

The trial will also compare arthroscopic capsuloligamentous repair (Bankart + Remplissage Procedure) vs. coracoid transfer (Latarjet procedure) on:

1. Rates of recurrent shoulder dislocations and symptoms of instability up to 24 months' post- surgery;
2. Clinical outcomes measured by Western Ontario Shoulder Instability (WOSI) Index, American Shoulder and Elbow Society (ASES) score;
3. Physical examination: range of motion, strength, stability;
4. Return to previous level of activity;
5. Rate of shoulder-related complications and serious adverse events.

Study Design:

The investigators propose a multi-center pilot Randomized Clinical Trial of 82 patients across Canada, United States and Europe to compare the effect of capsuloligamentous repair (Bankart + Remplissage procedure) and coracoid transfer (Latarjet procedure) in patients with post-traumatic recurrent anterior dislocation. Eligible and consenting participants will be followed-up by the site for 24 months. Outcomes will be assessed at 2 weeks, 3 months, 6 months, 12 months, and 24 months post-surgery. Eligible participants will be randomized to one of two treatment groups:

1. Arthroscopic capsuloligamentous repair (Bankart + Remplissage Procedure)
2. Open or Arthroscopic coracoid transfer (Latarjet Procedure)

Once participants have provided informed consent, baseline demographics, relevant medical history, and details regarding their diagnosis will be collected from the participant, the attending surgeon, their medical record and through physical examination. Participants will also complete The Western Ontario Shoulder Instability Index (WOSI) and he American Shoulder and Elbow Surgeons questionnaire (ASES) at the time of enrolment.

After surgery, surgical and peri-operative details will be collected from the attending surgeon and the participant's medical records. Adverse events occurring during the surgical procedure or perioperative period will also be documented.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-50 years;
* Diagnosis of post-traumatic recurrent anterior dislocation. This will require a minimum of 2 episodes of documented dislocations either by radiographic evidence or documented reduction of anterior shoulder dislocation as well as physical examination eliciting unwanted glenohumeral translation with reproduction of symptoms;
* Mild glenoid bone loss as defined on CT by standardized and reproducible best-fit circle technique (>10% but <20%);
* Provision of informed consent.

Exclusion Criteria:

* Patients with concomitant injuries (cuff tear);
* Previous shoulder surgery;
* Patients that will likely have problems, in the judgment of the investigators, with maintaining follow-up;
* Epilepsy;
* Patients who are or at risk of being incarcerated;
* Diagnosis of multidirectional instability;
* Cases involving litigation or workplace insurance claims (e.g. WSIB);
* Confirmed connective tissue disorder (Ehlers-Danlos, Marfans) or Beighton hypermobility score > 6.
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 10 months
  Number of patients recruited
Protocol Adherence | 2 years
  Number of errors in randomization
Follow-up | 2 years
  Proportion of participants followed at two years

SECONDARY OUTCOMES:
Rate of Recurrence | 2 years
  Rate of recurrent dislocation and symptomatic instability between patients randomized to (capsuloligamentous repair + remplissage) and those receiving open Latarjet procedure.
Clinical Outcome | 2 years
  Measured by Western Ontario Shoulder Instability (WOSI) Index
Clinical Outcome | 2 years
  Measured by American Shoulder and Elbow Society (ASES) score

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan M, Bedi A, Degen R, Warner J, Bhandari M; STABLE Investigators. A pilot multicenter randomized controlled trial comparing Bankart repair and remplissage with the Latarjet procedure in patients with subcritical bone loss (STABLE): study protocol. Pilot Feasibility Stud. 2022 Jan 31;8(1):20. doi: 10.1186/s40814-022-00987-4. PMID 35101120